CLINICAL TRIAL: NCT04042649
Title: The Effect of Environmental Intervention on Critically-ill Surgical Patients With Delirium
Brief Title: Environmental Intervention on Delirious Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, professor, Asan Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AsanMC-Delirium
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Delirium
Keywords: intensive care unit; critically ill patients; environmental intervention
MeSH Terms: conditions — Delirium | interventions — Milieu Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-intervention (No Intervention): Critically ill patients didn't provide environmental intervention (help sleep cycle, provide comfortable environment)
- post-intervention (Experimental): After providing environmental intervention for critically ill patients
  Interventions: Behavioral: environmental intervention

INTERVENTIONS:
Behavioral: environmental intervention — provide environmental intervention (help sleep cycle, provide comfortable environment)
  Arms: post-intervention

SUMMARY:
The implementation of environmental intervention program reduced the duration of delirium and length of stay at the ICU in critically-ill surgical patients.

DETAILED DESCRIPTION:
Purpose: Delirium occurs among patients in intensive care unit at high rates and increases the risk for morbidity and mortality. The purpose of this study is to investigate the effects of environmental interventions for the prevention of delirium.

Methods: A total of 192 patients who had been admitted to the surgical intensive care unit (SICU) in Asan Medical Center during the pre-intervention period (Jun 2013 to Oct 2013) and the post-intervention period (Jun 2014 to Oct 2014) was enrolled and prospective cohort study was done. The environmental intervention included cognitive assessment, providing orientation and comfortable environment, and a proper sleeping environment. The primary outcomes were the incidence rate of delirium, time of delirium onset, and the duration of delirium.

ELIGIBILITY:
Inclusion Criteria:

* with an age of 18 years or older
* who understood the purpose of this study and agreed to participate
* stayed in the SICU for a period of 48 hours or longer

Exclusion Criteria:

* who remained unresponsive [defined as the Richmond Agitation-Sedation Scale (RASS) less than -4]
* who could not measure Confusion Assessment Method (CAM-ICU) due to severe visual or hearing disturbance
* who had a history of severe psychiatric or neurologic deficit
* who required an isolation room due to transplantation or immunologic compromise
* who were discharged from ICU within 48 hours
* who were re-admitted to the ICU
* who were less than 18 years old
* who were admitted to the Surgical ICU through another ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
the incidence rate of delirium | 5 month
time to delirium onset | 5 month
the duration of delirium | 5 month

SECONDARY OUTCOMES:
the number of days of ventilator use | 5 month
the length of stay at the SICU | 5 month
the length of stay at hospital | 5 month
the rate of re-admission to the SICU | 5 month
mortality rate. | 5 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hakjae Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Inouye SK. The dilemma of delirium: clinical and research controversies regarding diagnosis and evaluation of delirium in hospitalized elderly medical patients. Am J Med. 1994 Sep;97(3):278-88. doi: 10.1016/0002-9343(94)90011-6. PMID 8092177
- [Result] Holt R, Young J, Heseltine D. Effectiveness of a multi-component intervention to reduce delirium incidence in elderly care wards. Age Ageing. 2013 Nov;42(6):721-7. doi: 10.1093/ageing/aft120. Epub 2013 Aug 26. PMID 23978407
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] Arenson BG, MacDonald LA, Grocott HP, Hiebert BM, Arora RC. Effect of intensive care unit environment on in-hospital delirium after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Jul;146(1):172-8. doi: 10.1016/j.jtcvs.2012.12.042. Epub 2013 Jan 11. PMID 23317943